CLINICAL TRIAL: NCT06115876
Title: Kuwait Adult Diabetes Epidemiological Multidisciplinary (KADEM) Program
Acronym: KADEM
Status: Recruiting | Type: Observational
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RAHM2019-030; RAHM2019-030 (Other: Kuwait Foundation for the Advancement of Sciences)
Record Dates: First submitted 2023-10-16; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus Type 2, Diabetes Mellitus Type 1; NAFLD - Nonalcoholic Fatty Liver Disease; PreDiabetes
Keywords: Prediabetes; Kuwait; KFAS; Dasman Diabetes Institute; Diabetes Prevention; NAFLD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Non-alcoholic Fatty Liver Disease; Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, PBMC, DNA,
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-Diabetes: Fasting Blood glucose ≥ and <7 5.6mmol/L ≥100 and<126 mg/dL HbA1C 5.7% to 6.4% 2hr Oral Glucose Tolerance Test (OGTT) ≥7.8 and <11.1 mmol/L ≥140 and<200 mg/dL
- Diabetes: Fasting Blood glucose 7 mmol/L (126mg/dL) or higher HbA1C 6.5% or higher 2hr Oral Glucose Tolerance Test (OGTT) 11.1 mmol/L (200 mg/dL) or higher

SUMMARY:
Kuwait and the Gulf Region lack large longitudinal studies that identify risk factors dictating the onset of prediabetes and the progression to diabetes. The Kuwait Diabetes Epidemiology Program (KDEP), previously carried out at Dasman Diabetes Institute, was designed to develop a research dataset providing a random sampling of the Kuwaiti population. The dataset contained primarily epidemiology data for healthy, prediabetic and diabetic individuals; and was designed to serve as a resource for research and prevention programs on obesity, diabetes, and metabolic syndrome. The KDEP data supported research studies at DDI to delineate risk factors for metabolic disease from the views of genetics, biochemistry, immunology and epidemiology. One of the main limitations of the KDEP study was that it only captured a cross-sectional view of the participants in terms of diabetes status as well as lack of extensive phenotyping. In the current study, the investigators aim to perform a follow up on the non-diabetic KDEP cohort participants to enrich it with detailed physiological, genetic, biochemical and environmental data and thereby to establish an association between the development of diabetes and multidimensional risk factors. the investigatorswill also recruit family members of the KDEP and RA2010-005 participants as well as others with family history of diabetes to better identify familial patterns in risk factors. The outcome of this effort will immediately serve as a scientific baseline for developing prevention strategies for the control and management of obesity, diabetes and associated complications such as cardiovascular disease. Given the magnitude of the social and economic burden of diabetes on the Kuwaiti population, longitudinal data from the KDEP Follow-up study should play an important role in establishing the incidence of T2D progression in non-diabetic participants that were enrolled in the initial study as well as of progression to diabetes complications. This will have a positive impact on the population by providing clinicians with data to better target their patient management and by supporting policy and decision-makers in developing comprehensive health promotion programs to control these diseases at the national level.

DETAILED DESCRIPTION:
The rapid increase of obesity and the detrimental complications associated with it, particularly insulin resistance, Type 2 diabetes (T2D), hypertension and cardiovascular disorders, represent a major threat to public health. Epidemiological data from Arabian Gulf countries warned of the high prevalence of obesity and T2D 1-4. According to the International Diabetes Federation (IDF), Gulf States such as Bahrain, Kuwait, Oman, Saudi Arabia, and United Arab Emirates ranked amongst the 10 countries in the world with highest prevalence of T2D 2,4. It is also known that the effect of obesity on the risk of developing these disorders differs by ethnicity 5 for example, South Asians have a higher risk for hypertension, T2D, cholesterol profiles and cardiovascular disease 6. In Arab populations, high familial aggregation of diabetes and related disorders have been observed. The population is characterised by consanguineous marriages and large family size. The large number of T2DM genetic loci identified globally to date were derived using unrelated subjects as study cohorts and explains only a relatively small proportion of observed heritability (familial clustering) of T2DM 7. Possible explanations for the "missing heritability" may originate from the role of rare variants, copy number variants, and more complex rearrangements, gene-environment interactions and epigenetics 8,9. Family-based designs allow the segregation of rare variants in a pedigree; multiple copies of such rare variants facilitate the detection of their effects. Family-based studies require fewer samples than population-based studies and offer advantages in terms of quality control, robustness to population stratification, and uniformity in exposure to environmental factors (gene-environment interactions and epigenetics) or lineage-specific diseases that have pleiotropic effect on diabetes. They also offer the potential to combine linkage and association data. Arab populations, which often have a high rate of consanguinity 10, offer a large potential for family-based designs as they show familial gene clustering for diabetes and metabolic traits 11-13. However, except for few studies, such as the "Oman Family Study" 14 and a study on an extended family from the UAE, no notable familial study for diabetes risk loci has been reported for the Arab population. Both the above-mentioned studies confirmed well-established gene loci but failed to identify any novel "rare" variants.

Paralleling this world-wide increase in obesity is the increase in the incidence and prevalence of non-alcoholic fatty liver disease (NAFLD). The global prevalence of NAFLD is about 24% whereas its prevalence in the Middle East Region is more than 30% 15. Given the high percentage of obesity in a country like Kuwait, the prevalence of NAFLD would be expected to be much higher as well. Hepatic steatosis is the underlying manifestation of NAFLD and is clinically defined as a hepatic triglyceride content that exceeds 5%. Even though NAFLD was considered a benign manifestation, it is currently clear that it is linked to the development of steatohepatitis, fibrosis, cirrhosis and eventually the development of hepatocellular carcinoma 16.

Liver lipid content is regulated by an intricate equilibrium between lipid uptake and secretion. The main sources for hepatic lipids are adipose tissue lipolysis (which is the source of about 60% of liver triglyceride), dietary intake and de novo lipogenesis. On the other hand, hepatic lipid content can be reduced by lipid secretion (primarily VLDL secretion) and mitochondrial fatty acid oxidation. High-fat and glucose diets as well as obesity and insulin resistance lead to increased influx of fat into the liver and the accumulation of intracellular triglyceride in hepatic tissues and ultimately to the development of nonalcoholic steatohepatitis (NASH).

Kuwait and the Gulf Region lack large longitudinal studies to identify risk factors for the progression of metabolic dysfunction that leads to the transition from prediabetes to diabetes. The Kuwait Diabetes Epidemiology Program (KDEP) (RA-2010-004) was designed to develop a research dataset which offers a full characterization of the Kuwaiti population and contains detailed clinical, genetic, immunological, physiological, biochemical and environmental data which can serve as a resource for future research and prevention programs to fight against obesity, diabetes, and metabolic syndrome. A number of papers have been published from the original cross-sectional study reporting data regarding the studied population such as the prevalence of cardiovascular disease risk factors in South Asian expatriates in Kuwait 17, the association between adipokines and hsCRP and the Metabolic Syndrome in Arabs as well as ghrelin and adiponectin in Arabs 18-20. Another paper looked at vitamin D levels in Arab and Asians 21. Two additional studies performed genome-wide genotyping of the study cohort, resulting in papers that reported genetic risk loci for metabolic traits 22,23. An eighth paper characterizes a novel biomarker called betatrophin, showing that betatrophin levels in T2D was increased compared to non-diabetic participants. Betatrophin levels showed significant increase in subjects with longer duration of T2D 24. A major limitation of these studies is the cross-sectional design that could not support relationships between the cause and effect.

In the current study, the investigators aim to do a follow up on the KDEP to provide datasets to support development of evidence-based optimal prevention strategies for the control and management of obesity and its complications, including diabetes and cardiovascular disease. Data collected in the KDEP Follow-up study will also support policy and decision-makers in implementing comprehensive health promotion programs to control these diseases at the national level and to establish their appropriateness and cost effectiveness for the whole population. The outcome of this effort will immediately serve as a database for genetic and biochemical risk factors as well as it will provide data that can be used to potentially establish risk scoring based on regional data that is applicable to the Arab population and other people living in Kuwait. It will also support efforts that implement comprehensive health promotion programs to prevent and manage these diseases at the national level. Given the magnitude of the human and the economic burden of diabetes on the Kuwaiti population, longitudinal data from the KDEP Follow-up study should contribute to reducing the impact of diabetes and related metabolic complications on the population as well as expanding the original cohort. It will also act as a guide to assist health policy and decision makers in their planning strategies for adapting appropriate preventive measures.

Study Rationale

The primary aim of the present study is to recall all 3970 non-diabetic participants in KDEP as well as other high risk individuals and determine the incidence of prediabetes and new onset T2DM using a 75-gram OGTT according to the ADA criteria. the investigators also will determine the incidence of microvascular (i.e. retinopathy, nephropathy, and neuropathy) and macrovascular complications in subjects who converted to T2DM and those with prediabetes compared to NGT subjects. the investigators also will perform detailed biochemical/molecular workup to identify risk factors associated with the progression to prediabetes/T2DM and associated with the development of vascular (micro- and macrovascular) complications.

the investigators will also do OGTT/ Hyperglycemia CLAMP (H-CLAMP) and Euglycemic Clamp for a subset of (250) participant.

Objectives

The primary objective of the study is to determine the incidence of T2DM and its complications in Kuwaiti population. the investigators also will identify risk factors associated with the development of T2DM and/or its vascular complications. Therefore, the investigators propose the following SPECIFIC AIMS:

Specific Aim 1: Determine the 4-7 year incidence rate of T2DM in KDEP cohort according to the ADA criteria.

Specific Aim 2: Determine the incidence rate of microvascular (retinopathy, nephropathy and neuropathy) and macrovascular diabetic complications in subjects with prediabetes and new onset diabetes in KDEP cohort.

Specific Aim 3: Identify metabolic/biochemical/molecular factors associated with the development of diabetes and its vascular complications in KDEP cohort.

ELIGIBILITY:
Inclusion Criteria:

People who participated in the original KDEP study. People with prediabetes. Type 2 Diabetes patients.

Exclusion Criteria:

People are unwilling to sign the consent form. Pregnant women.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be performed in several phases. At the first phase we will recall subjects with prediabetes (n=1787), because we anticipate that many of whom have converted to T2DM. Other high risk individuals will be also enrolled in study for OGTT assessment. Additionally, subjects who are already diagnosed with diabetes (T1DM and / or T2DM) and/or receive antidiabetic therapy & participants between age of 10 and 21 years will not receive an OGTT. They only will receive a single blood draw (at baseline), and complete the questionnaire and all other imaging measurements described above.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2027-05-23 (Estimated); Study Completion 2027-05-23 (Estimated)

PRIMARY OUTCOMES:
Conversion to Diabetes | 5 years
  The investigators will monitor using HbA1C and FPG or 2-hr plasma glucose to diagnose new cases of diabetes in the original cohort. Type 2 Diabetes will be diagnosed according to ADA criteria.
Conversion to Pre-Diabetes | 5 years
  The investigators will monitor using HbA1C and FPG or 2-hr plasma glucose the conversion from normoglycemia to prediabetes in the original cohort. Pre-diabetes will be diagnosed according to ADA criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared after proper agreement plans
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: mid-2024 till 2027
URL: https://www.dasmaninstitute.org/ddi-launches-a-new-study-the-kuwait-adult-diabetes-epidemiological-multidisciplinary-or-kadem/